CLINICAL TRIAL: NCT07149870
Title: Pain Management Teams Using Whole Health to Optimize Function and Safety in Veterans: The TEAMWORK Trial
Acronym: TEAMWORK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDR 24-122; 1UG3AT012256-01A1 (Other Grant/Funding Number: VA-HSR (VA Health Systems Research))
Record Dates: First submitted 2025-08-06; First posted 2025-09-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
Keywords: Opioid Use; Opioid Safety; Pain; Chronic Pain; Long-term Opioid Therapy; Pain Management; Opioid; Whole Health; Coaching; Whole Health Coaching; Pain, Chronic; Buprenorphine
MeSH Terms: conditions — Chronic Pain; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: The interventional component of this trial includes 2 arms: 1) Pain management team usual care; and 2) Pain management team usual care with a Whole Health coach. Participants are randomized 1:1 at the individual level.
  The intervention model adds to the existing approach by enhancing Pain management teams (PMTs) with Whole Health coaching. Coaches use the VA Whole Health Personalized Health Planning and Coaching approach to promote wellness in Veterans with chronic pain.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not know participant assignment at 1-, 3-, 6-, and 12-month assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PMT-WHC (Experimental): The PMT-WHC group will receive PMT Usual Care plus 8 sessions of Whole Health Coaching (WHC)
  Interventions: Other: Pain Management Team + Whole Health Coach (PMT-WHC); Other: Pain Management Team-Usual Care (PMT-UC)
- PMT-UC (Active Comparator): The PMT-UC group will receive PMT Usual Care
  Interventions: Other: Pain Management Team-Usual Care (PMT-UC)

INTERVENTIONS:
Other: Pain Management Team + Whole Health Coach (PMT-WHC) — Whole Health Coaching (WHC) begins by completing a Personalized Health Inventory (PHI), where progress is evaluated within 8 dimensions of health and wellness. The PHI culminates in defining personal values and overall goals for health and wellness (i.e., "What do you want your health for?"). This is used to create goals for a Personal Health Plan. The Plan emphasizes self-management strategies to manage pain. After the Plan is developed, ongoing support is provided from the Coach through 8 coaching sessions over approximately 5 months.
  Other Names: PMT-WHC
  Arms: PMT-WHC
Other: Pain Management Team-Usual Care (PMT-UC) — Pain Management Team-Usual Care (PMT-UC) involves working with VA PMTs that includes working with PMTs comply with legislation requiring each medical center to have PMTs with expertise in pain, addiction, behavioral approaches, and rehabilitation approaches. PMTs will conduct multidisciplinary intakes (at least two provider types) with biopsychosocial assessments for all new patients. Follow-up care will be determined by the PMTs based on what is clinically indicated (with recommended minimum medication management follow ups at 1- 3- and 6-months for patients making medication changes).
  Other Names: PMT-UC

SUMMARY:
The focus of this study is to determine whether adding Whole Health Coaching (WHC) improves pain care among adults with chronic pain and who are currently working with a pain management team (PMT) at the VA.

DETAILED DESCRIPTION:
This multisite pragmatic effectiveness-implementation hybrid type 2 trial will randomize 432 patients to compare Pain Management Team - Usual Care (PMT-UC) vs. Pain Management Team Usual Care + Whole Health Coaching (PMT-WHC) on the primary composite outcome of pain-related interference and opioid safety. The investigators will also evaluate the impact of PMT-WHC on buprenorphine initiation and maintenance, evaluate implementation facilitation strategies for building and sustaining PMTs, and conduct a budget impact analysis.

The primary study goal is to evaluate the effectiveness of adding Whole Health Coaching to PMTs adhering to VA standards on the primary composite outcome of pain-related function and opioid safety, and secondary outcomes of wellbeing and physical functioning. Participants will have a 50/50 random chance of being assigned to (a) continuing to receive usual care from the PMT or (b) (a) receiving WHC in addition to the usual care provided by the PMT.

Both groups will receive usual care from the PMT, which will include a baseline evaluation with at least two PMT clinicians. Follow-up appointments will vary based on clinical judgment of the PMT members, but most patients will be followed for at least six months with at least three follow-up appointments. Both groups will complete questionnaires via telephone at (1) baseline, (2) month 1, (3) month 3, (4) month 6, and (5) month 12. The questionnaires will ask about personal characteristics and demographics, pain, physical function, ability to do activities, social support, sleep, mental health, use of medications and health services, and substance use.

If assigned to participate in PMT-WHC, participants will work with a Whole Health Coach for eight (8) individual sessions. Whole Health Coaching begins by completing a Personalized Health Inventory (PHI), where progress is assessed within eight (8) dimensions of health and wellness: Physical, Emotional, Social, Spiritual, Intellectual, Environmental, Financial, and Occupational health. The Inventory culminates in defining personal values and overall goals for health and wellness (i.e., "What do you want your health for?") based on a person's mission, aspiration, and purpose. This will be used to create goals that become part of a Personal Health Plan. The Personal Health Plan emphasizes self-management strategies to manage pain. After the Plan is developed, ongoing support is provided from the Coach in coaching sessions. Coaches will meet with participants on a biweekly basis for the first three (3) months after randomization and on a monthly basis for the final two (2) months, for a total of eight (8) sessions across approximately five (5) months. The sessions with the WHC will be recorded (audio recordings only, no photographs or video recordings). However, participation is still available in this study if participants decline to be recorded.

Participants may also be selected to participate in a qualitative interview. If selected, the interview covers participant experiences and opinions about working with the PMT, and, if relevant, the WHC. This interview will be recorded and will be approximately 60 minutes. Participants are not required to complete the interview and are still eligible to participate in this research study if the interview portion is declined.

The study will also evaluate implementation facilitation as a strategy to support PMTs in implementing care for patients with pain and opioid safety concerns. Implementation facilitation will include audit and feedback and other strategies tailored to each site. A budget impact analysis will monitor implementation and intervention costs.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA:

1. High-impact chronic pain (defined using the Graded Chronic Pain Scale - Revised).

   -AND-
2. Active prescription for LTOT (>90 days continuous prescription). -AND-
3. Exhibit evidence of at least ONE opioid safety concern (*indicators of opioid safety concerns described below).

   * Opioid safety concerns for inclusion purposes include:

     1. moderate-to-high dose opioid prescription (morphine equivalent daily dose >60mg)
     2. comorbid conditions that increase the risk of opioids including chronic pulmonary disease (e.g., emphysema, chronic bronchitis, asthma, or other breathing problems), sleep apnea, chronic kidney disease, chronic hepatitis or cirrhosis
     3. active high-risk co-prescriptions, including benzodiazepine prescription (any dose of long-term treatment), gabapentin prescription (1800mg or higher) or pregabalin prescription (150mg or higher)
     4. risk of substance use and/or potential opioid misuse as evidenced by unexpected urine toxicology findings in past 6-months OR any documented active substance use disorder (other than tobacco or caffeine) as evidenced by at least 2 encounters within the previous 12-months with a substance use disorder diagnosis.
     5. a positive TAPS score
     6. a positive AUDIT-C score
     7. presence of any adverse events as measured by the adverse effects checklist administered during screening
     8. reported score of >8 as measured by the Prescribed Opioids Difficulties Scale (PODS).

Exclusion Criteria:

1. Moderate to severe cognitive impairment as measured by the Blessed Orientation Memory Concentration (BOMC) screening tool.

   -OR-
2. Current/active prescription for buprenorphine or receipt of buprenorphine in the previous 6-months.

   -OR-
3. Inability to read or understand English. -OR-
4. Severely impaired hearing or speech that would preclude participation in telephone interviews or appointments with the Whole Health Coach.

   -OR-
5. Terminal illness/disease with a prognosis of <12 months. -OR-
6. Planned move/relocation outside of the treatment areas of the participating enrolling study sites.

   -OR-
7. Participants actively working with a Whole Health Coach or who have worked with a Whole Health Coach in the 6-months prior to enrollment.

   -OR-
8. Major surgical procedure planned during the study treatment or follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite of Pain Interference and Opioid Safety | 6 months
  The primary outcome for the clinical trial is a composite of pain-related interference and opioid safety where success at the individual level is only met when pain-related interference and opioid safety improve. The pain component of the composite primary outcome, measured at 6-month follow-up, will be change in pain interference from baseline, measured on the Brief Pain Inventory - Interference scale, categorized as improved/not improved with improvement defined as a ≥1 point reduction in pain-related interference. The opioid safety component of the composite primary outcome will be defined as success in one or more of the following: (1) initiating and continuing buprenorphine for at least 90 days, or (2) evidence of an opioid taper (i.e., a >25% reduction in daily full agonist opioid dose, including opioid discontinuation), at 6 months.

SECONDARY OUTCOMES:
Opioid Safety | 6 months, 12 months
  We will look at a more expansive list of indicators of improved opioid safety as a secondary outcome, including: (1) initiating and continuing buprenorphine for at least 90 days, (2) evidence of an opioid taper (i.e., a >25% reduction in daily full agonist opioid dose, including opioid discontinuation), (3) 25% reduction in gabapentin dose, (4) 25% reduction in benzodiazepine dose, (5) resolution of a positive baseline TAPS-2 score, (6) resolution of a positive AUDIT-C score, (7) reduction in opioid-related difficulties as measured by the Prescribed Opioids Difficulties (PODS) scale, and (8) reductions in sleepiness as measured by the Epworth Sleepiness Scale.
Well-Being Signs (WBS) Tool | 6 months, 12 months
  The Wellbeing Signs Tool is a three (3) item screening tool with items asking respondents to rate how well they are doing in their daily lives; higher scores indicated better wellbeing and life satisfaction.
Pain Interference | 6 months, 12 months
  The pain component of the composite primary outcome, measured at 6-month follow-up, will be change in pain interference from baseline, measured on the Brief Pain Inventory - Interference scale, categorized as improved/not improved with improvement defined as a ≥1 point reduction in pain-related interference.
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Short Form 6b | 6 months, 12 months
  Physical Functioning: An assessment of the impact of pain on several aspects of functioning, including social and emotional processes as well as physical function (e.g., how much did pain interfere with your day to day activities).
Composite of Pain Interference and Opioid Safety | 12 months
  We will examine the composite of pain-related interference and opioid safety (primary outcome at 6 months) as a secondary outcome for durability of effects at 12 months. The pain component of the composite primary outcome, measured at 12-month follow-up, will be change in pain interference from baseline, measured on the Brief Pain Inventory - Interference scale, categorized as improved/not improved with improvement defined as a ≥1 point reduction in pain-related interference. The opioid safety component of the composite primary outcome will be defined as success in one or more of the following: (1) initiating and continuing buprenorphine for at least 90 days, or (2) evidence of an opioid taper (i.e., a >25% reduction in daily full agonist opioid dose, including opioid discontinuation), at 12 months.

OTHER OUTCOMES:
World Health Organization - Quality of Life (WHOQOL- 2) | 6 months, 12 months
  The WHOQOL assesses individuals' perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. The 2-item version of this measure (recommended by the NIH HEAL CDE Initiative) will be used.
Patients' Global Impression of Change (PGIC) | 6 months, 12 months
  Global Satisfaction with Treatment: A scale for respondents to rate the level of change experienced following treatment. The PGIC is a 7-point scale from 1 (very much better) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Edmond, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Karen H Seal, MD MPH, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (5):
- United States (5):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Central Arkansas Veterans Healthcare System , Little Rock, AR, Little Rock, Arkansas
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Boise VA Medical Center, Boise, ID, Boise, Idaho

IPD SHARING:
Plan to Share IPD: No